CLINICAL TRIAL: NCT02915042
Title: A Randomized, Double-Blinded, Placebo Controlled Trial Using Single Dose Dexmedetomidine In The Treatment Of Pain In Patients Undergoing Cleft Palate Repair
Brief Title: Dexmedetomidine vs Placebo for Pediatric Cleft Palate Repair
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment concerns
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Chris Glover, Dr. Chris Darrel Glover Assistant Professor Anesthesiology Texas Children's Hospital Baylor College of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-34431
Record Dates: First submitted 2016-09-23; First posted 2016-09-26 (Estimated); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Cleft Palate
Keywords: Pain; dexmedetomidine; postoperative
MeSH Terms: conditions — Cleft Palate; Pain | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Intervention group 1: pre-operative administration of IV dexmedetomidine 1mcg/kg
  Interventions: Drug: Dexmedetomidine
- Placebo group (Placebo Comparator): Intervention group 2: placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — Analgesic Efficacy
  Other Names: Precedex
  Arms: Experimental group
Drug: Placebo — Saline placebo
  Other Names: Saline
  Arms: Placebo group

SUMMARY:
The primary objective of this study is to evaluate the efficacy of administering intravenous dexmedetomidine as a single preemptive dose to placebo in reducing the total 24 hour dose of opioids as measured on a weight adjusted morphine equivalent basis.

DETAILED DESCRIPTION:
The eligibility of the patient to participate in this study will be determined by the Investigator on the basis of the inclusion and exclusion criteria. Consent will be obtained from eligible patients only.

The following is the standard intraoperative anesthesia protocol utilized at Texas Children's Hospital for all children undergoing this procedure of cleft palate repair even if they are not part of the study: (1) Induction of anesthesia via a face mask with sevoflurane 6-8% and 70% N2O / 30% O2 (2) A peripheral IV will be inserted and glycopyrrolate 5-10 mcg/kg IV administered to dry oral secretions and reduce vagal responses. (3) Tracheal intubation using appropriate equipment in keeping with the clinical judgment of the anesthesia care provider. The protocol will permit the administration of propofol up to 3 mg/kg over 20-30 seconds to increase the depth of anesthesia prior to tracheal intubation if the Attending Anesthesiologist deems it necessary. (4) General anesthesia maintained with Sevoflurane/isoflurane with inhaled concentrations adjusted to keep blood pressure and heart rates within 20% of baseline. (5) Nitrous oxide will be discontinued and the lowest inspired oxygen concentration will be administered to reduce risks of airway fires while avoiding hypoxemia. (6) Fentanyl 1-2 mcg/kg administered at the start of the procedure with subsequent fentanyl 1 mcg/kg boluses as needed if the heart rate and blood pressure are increased per vital signs (HR and BP) variance greater than 20% of baseline (7) Dexamethasone 0.5 mg/kg IV. (8) Rocuronium 0.6 -1 mg/kg IV may be administered for paralysis if this is clinically indicated in the opinion of the Attending Anesthesiologist. (9) Local infiltration with 0.5% lidocaine with 1:200,000 epinephrine will be administered by the surgeon at the site of the palatoplasty in keeping with our current surgeon practice. (10) Ondansetron 0.1 mg/kg IV at the end of the procedure (11) Anesthetic gases will be discontinued at the end of the procedure and 100% oxygen administered prior to tracheal extubation. If rocuronium was used neuromuscular blockade will be antagonized with neostigmine 0.07 mg/kg and glycopyrrolate 10 mcg/kg. The timing of tracheal extubation will be based on clinical indications and the judgment of the Attending Anesthesiologist.

The above standardized management will be followed for all children undergoing this operation even if they are not part of the study. The experimental part of the protocol will involve randomization of subjects in a 1:1 ratio to receive intravenous dexmedetomidine or placebo. Randomization will occur by the pharmacy using a computer generated random number. The study will be double-blind with respect to the treatment assignment. The investigational pharmacy will mix and deliver either dexmedetomidine 1 mcg/kg in a concentration of 4 mcg/ml or placebo to the anesthesia provider on the day of surgery. The assigned study drug will be administered when the heart rate and blood pressure have returned to acceptable stable levels after tracheal intubation and before the surgeon has started the palatal injection of lidocaine with epinephrine. Placebo or dexmedetomidine will be administered in a similar fashion as an IV infusion over 10 minutes as recommended to avoid bradycardia,hypertension, hypotension or other cardiac events. . Persistent bradycardia (greater than 30% reduction from baseline for more than 1 minute) will be managed with administration of atropine 0.01 mg/kg. An immediate rise in blood pressure will be treated with an increase in the inspired concentration of inhaled anesthetics. If there is hypertension (greater than 30% rise in value from baseline), the inspired concentration of inhaled anesthetics will be increased. Persistent hypotension (greater than 30% decrease from baseline levels for more than 1 minute) will be treated with fluid bolus of 5-10 ml/kg and decreasing the concentration of the volatile anesthetic. Other drugs may be used in keeping with the clinical judgment of the Attending Anesthesiologist.

Postoperative management will not be changed for the purposes of the study. In keeping with standard practices in the TCH, all patients in the PACU will be monitored with continuous pulse oximetry, EKG and serial non-invasive blood pressure measurements. Pain will be assessed using an age appropriate observational scale- the FLACC score for younger patients and the FACES score for older co-operative patients. Pain scores are recorded on arrival to the PACU, when awake and at 30 minute intervals. If the FLACC score is greater than 4 or the FACES greater than 2, patients will receive morphine 25 mcg/kg IV to be repeated as required in 10 minutes if adequate pain control has not been achieved. Supplemental oxygen will be administered till the child can maintain an oxygen saturation greater than 92% in room air. Emergence delirium will be determined using the PAED score and children with scores of greater than 12 will receive therapy in keeping with the clinical judgment of the Attending Anesthesiologist (additional opioids or IV propofol). The child will be discharged to the floor when awake, can maintain patency of the airway, have stable vital signs, a pain score less than 4 and an Aldrete score of at least 9.

Patients will be transferred to the floor where they will receive the current standard postoperative regimen used by our plastic surgery service care for this procedure. This will includeHycet 0.135mg/kg every 4 hours when needed. Morphine 0.025 mg/kg IV every 4 hours will be made available as a rescue analgesia for break through pain. Nurses record pain scores on the FLACC or FACES scale depending on the age of the patient and ability to cooperate. Rescue analgesia will be provided based on a nursing assessment that the pain is poorly controlled (FLACC score greater than 4 or FACES score greater than 2) after receiving oral pain medications. Non -steroidal anti-inflammatory drugs are usually avoided in these children because of concerns for bleeding from the raw mucosal surfaces at the site of the surgery.

We will record all perioperative, intraoperative and postoperative drugs administered to patients, pain scores, Pediatric Anesthesia Emergence Delirium (PAED) scores in the PACU, pain scores and rescue medications administered during the stay in the PACU and on the floor. The time to first rescue medication, oral intake, and discharge from the PACU and the hospital will also be recorded along with adverse events such as vomiting, constipation, pruritis, agitation, respiratory depression or excessive sedation. Any interventions to treat these will be noted.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 6mo to 8 years of age scheduled to undergo primary or secondary cleft repair.

Exclusion Criteria:

* Patients with significant cognitive impairment
* Patients with various syndromes known to be associated with difficult airways(e.g. Goldenhar's syndrome, Treacher- Collins, Trisomy 13 or 18, Pierre Robin, etc.)
* Have a prior history of allergy, hypersensitivity or contraindication to any drug used for anesthesia including opioids (morphine, fentanyl, hydrocodone) and inhalation agents(i.e. children with susceptibility to malignant hyperthermia)
* Have a history of congenital bleeding diathesis(e.g. hemophilia) or any active clinically significant bleeding, impaired renal or hepatic function
* Children with heart failure, heart block, ventricular dysfunction, cardiomyopathy, myocarditis or congenital heart disease where cardiac output is rate dependent and relies on A-V synchrony (e.g. single ventricle). Children with well controlled atrial or ventricular septal defects, patent ductus arteriosus, repaired coarctation of the aorta will qualify if they have no cardiac rhythm or hypertension problems.
* Children with uncontrolled hypertension, intracranial vascular malformations, Moya Moya disease or intracranial hypertension.
* Any child who has received an investigational drugs within 30 days before study drug administration.
* Inability of the parent or legal guardian to understand the requirements of the study or be unwilling to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board) and agree to abide by the study restrictions.
* Be otherwise unsuitable for the study, in the opinion of the Investigator.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2017-12-31 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain control | 24 hours
  Assessment of and clinical measurement that one treatment group will be better with postoperative pain management than the non-treatment group, which would be similar to published data for children undergoing this procedure. This will be measured in a mean pain score. There will be integrating of pain scores and morphine consumption.
Opioid consumption | 24 hours
  Opioid consumption is measured in mean morphine equivalent dose in mcg/kg, this will be integrated with the pain scores.

SECONDARY OUTCOMES:
The number of children with FLACC scores greater than 4 | 24 hours
  FLACC Pain Scores
Time to first rescue analgesia | 24 hours
  Time in minutes to administration of first dose of rescue analgesia
Respiratory depression | 24 hours
  Patients with SPO2 less than 85%
Postoperative vomiting | 24 hours
  postoperative emesis

CONTACTS AND LOCATIONS:
Overall Officials: Chris D. Glover, MD, Principal Investigator — Baylor College of Medicine - Texas Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelly LE, Rieder M, van den Anker J, Malkin B, Ross C, Neely MN, Carleton B, Hayden MR, Madadi P, Koren G. More codeine fatalities after tonsillectomy in North American children. Pediatrics. 2012 May;129(5):e1343-7. doi: 10.1542/peds.2011-2538. Epub 2012 Apr 9. PMID 22492761
- [Background] Mason KP, Lerman J. Review article: Dexmedetomidine in children: current knowledge and future applications. Anesth Analg. 2011 Nov;113(5):1129-42. doi: 10.1213/ANE.0b013e31822b8629. Epub 2011 Aug 4. PMID 21821507
- [Background] Pickard A, Davies P, Birnie K, Beringer R. Systematic review and meta-analysis of the effect of intraoperative alpha(2)-adrenergic agonists on postoperative behaviour in children. Br J Anaesth. 2014 Jun;112(6):982-90. doi: 10.1093/bja/aeu093. Epub 2014 Apr 11. PMID 24727829
- [Background] Sun Y, Lu Y, Huang Y, Jiang H. Is dexmedetomidine superior to midazolam as a premedication in children? A meta-analysis of randomized controlled trials. Paediatr Anaesth. 2014 Aug;24(8):863-74. doi: 10.1111/pan.12391. Epub 2014 Mar 26. PMID 24666837
- [Background] Schnabel A, Reichl SU, Poepping DM, Kranke P, Pogatzki-Zahn EM, Zahn PK. Efficacy and safety of intraoperative dexmedetomidine for acute postoperative pain in children: a meta-analysis of randomized controlled trials. Paediatr Anaesth. 2013 Feb;23(2):170-9. doi: 10.1111/pan.12030. Epub 2012 Oct 9. PMID 23043461
- [Background] Olutoye OA, Glover CD, Diefenderfer JW, McGilberry M, Wyatt MM, Larrier DR, Friedman EM, Watcha MF. The effect of intraoperative dexmedetomidine on postoperative analgesia and sedation in pediatric patients undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Aug;111(2):490-5. doi: 10.1213/ANE.0b013e3181e33429. Epub 2010 Jul 7. PMID 20610555
- [Background] Petroz GC, Sikich N, James M, van Dyk H, Shafer SL, Schily M, Lerman J. A phase I, two-center study of the pharmacokinetics and pharmacodynamics of dexmedetomidine in children. Anesthesiology. 2006 Dec;105(6):1098-110. doi: 10.1097/00000542-200612000-00009. PMID 17122572
- [Background] Potts AL, Anderson BJ, Warman GR, Lerman J, Diaz SM, Vilo S. Dexmedetomidine pharmacokinetics in pediatric intensive care--a pooled analysis. Paediatr Anaesth. 2009 Nov;19(11):1119-29. doi: 10.1111/j.1460-9592.2009.03133.x. Epub 2009 Aug 25. PMID 19708909
- [Background] Mason KP, Robinson F, Fontaine P, Prescilla R. Dexmedetomidine offers an option for safe and effective sedation for nuclear medicine imaging in children. Radiology. 2013 Jun;267(3):911-7. doi: 10.1148/radiol.13121232. Epub 2013 Feb 28. PMID 23449958
- [Background] Tobias JD, Gupta P, Naguib A, Yates AR. Dexmedetomidine: applications for the pediatric patient with congenital heart disease. Pediatr Cardiol. 2011 Dec;32(8):1075-87. doi: 10.1007/s00246-011-0092-8. Epub 2011 Sep 10. PMID 21909772
- [Background] Chen ZF, Chen YK, Guo Y, Jiang H. [Effect of dexmedetomidine on emergence agitation after oral and maxillofacial surgery]. Shanghai Kou Qiang Yi Xue. 2013 Dec;22(6):698-701. Chinese. PMID 24469137
- [Background] Patel A, Davidson M, Tran MC, Quraishi H, Schoenberg C, Sant M, Lin A, Sun X. Dexmedetomidine infusion for analgesia and prevention of emergence agitation in children with obstructive sleep apnea syndrome undergoing tonsillectomy and adenoidectomy. Anesth Analg. 2010 Oct;111(4):1004-10. doi: 10.1213/ANE.0b013e3181ee82fa. Epub 2010 Aug 12. PMID 20705788
- [Background] Nour C, Ratsiu J, Singh N, Mason L, Ray A, Martin M, Hassanian M, Uhler J, Applegate RL 2nd. Analgesic effectiveness of acetaminophen for primary cleft palate repair in young children: a randomized placebo controlled trial. Paediatr Anaesth. 2014 Jun;24(6):574-81. doi: 10.1111/pan.12393. Epub 2014 Apr 2. PMID 24697925
- [Background] Kayyal TA, Wolfswinkel EM, Weathers WM, Capehart SJ, Monson LA, Buchanan EP, Glover CD. Treatment effects of dexmedetomidine and ketamine on postoperative analgesia after cleft palate repair. Craniomaxillofac Trauma Reconstr. 2014 Jun;7(2):131-8. doi: 10.1055/s-0034-1371446. Epub 2014 Feb 28. PMID 25045418
- [Background] Berde CB, Sethna NF. Analgesics for the treatment of pain in children. N Engl J Med. 2002 Oct 3;347(14):1094-103. doi: 10.1056/NEJMra012626. No abstract available. PMID 12362012
- [Background] Lonnqvist PA, Morton NS. Postoperative analgesia in infants and children. Br J Anaesth. 2005 Jul;95(1):59-68. doi: 10.1093/bja/aei065. Epub 2005 Jan 21. No abstract available. PMID 15668207
- [Background] Mason KP, Zurakowski D, Zgleszewski S, Prescilla R, Fontaine PJ, Dinardo JA. Incidence and predictors of hypertension during high-dose dexmedetomidine sedation for pediatric MRI. Paediatr Anaesth. 2010 Jun;20(6):516-23. doi: 10.1111/j.1460-9592.2010.03299.x. Epub 2010 Apr 14. PMID 20412458
- [Background] Mascha EJ, Turan A. Joint hypothesis testing and gatekeeping procedures for studies with multiple endpoints. Anesth Analg. 2012 Jun;114(6):1304-17. doi: 10.1213/ANE.0b013e3182504435. Epub 2012 May 3. PMID 22556210
- [Background] Dai F, Silverman DG, Chelly JE, Li J, Belfer I, Qin L. Integration of pain score and morphine consumption in analgesic clinical studies. J Pain. 2013 Aug;14(8):767-77.e8. doi: 10.1016/j.jpain.2013.04.004. Epub 2013 Jun 3. PMID 23743256
- [Background] Farag E, Atim A, Ghosh R, Bauer M, Sreenivasalu T, Kot M, Kurz A, Dalton JE, Mascha EJ, Mounir-Soliman L, Zaky S, Ali Sakr Esa W, Udeh BL, Barsoum W, Sessler DI. Comparison of three techniques for ultrasound-guided femoral nerve catheter insertion: a randomized, blinded trial. Anesthesiology. 2014 Aug;121(2):239-48. doi: 10.1097/ALN.0000000000000262. PMID 24758775
- See also: Medical staff resource — https://www.aspirus.org/for-providers